CLINICAL TRIAL: NCT06020391
Title: Cooperation Across Healthcare Service Levels for Medication Reviews in Older People with Polypharmacy Admitted to a Municipal In-patient Acute Care Unit (The COOP II Study): a Randomized Controlled Trial
Brief Title: Cooperation for Better Treatment of Polypharmacy in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); South-Eastern Norway Regional Health Authority (Other); City of Oslo (Unknown)
Responsible Party: Principal Investigator, Rita Romskaug, MD, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022066
Record Dates: First submitted 2023-08-22; First posted 2023-08-31 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Drug Usage
Keywords: Polypharmacy; Geriatrics; Drug review; Medication review; Elderly

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Collaborative drug review.
  Interventions: Other: Collaborative drug review
- Control group (No Intervention): Usual care.

INTERVENTIONS:
Other: Collaborative drug review — 1. Structured, clinical drug review including medical history, physical examination, and supplementary tests. The work-up will be aimed at evaluating whether current medications are indicated, whether the patient's medical conditions are satisfactorily compensated, whether dosages are appropriate, whether the patient has adverse drug effects, and whether drug-drug or drug-disease interactions are present or likely to occur. The MipAC physicians will receive clinical supervision from a consultant in geriatric medicine.
  2. The MipAC physician will offer the patient's FP a telephone meeting with the purpose of combining the assessments of the MipAC physician and the competence of the FP in a common drug review. The two physicians will review the patient's drug list systematically and discuss if any adjustments should be done, as well as the patient's need for further follow-up.
  Arms: Intervention group

SUMMARY:
The elderly population today relies heavily on medication consumption. While there are cases where using multiple medications is necessary and reasonable, it also increases the risk of inappropriate treatment and adverse drug effects. This randomized, controlled trial aims to examine the effectiveness of incorporating drug reviews as an integral part of clinical practice for older patients admitted to a Municipal in-patient acute care (MipAC) unit in Oslo, Norway. The intervention involves a clinical drug review conducted by a MipAC physician under the guidance of a geriatrician, followed by a telephone consultation between the MipAC physician and the patient's family physician (FP). The primary outcome measure is health-related quality of life, while secondary outcome measures include physical and cognitive function, dry mouth, hospital admissions, and survival. The environmental impact of the study intervention will also be assessed and compared to usual care.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of collaborative drug reviews by MipAC physicians, supervised by geriatricians, and FPs on clinically relevant outcome measures in the MipAC patient population aged 70+. The investigators will also assess the environmental impact of the study intervention and compare it to usual care.

The study is a randomized, single-blind, controlled trial with 16 weeks follow-up. In addition, we plan to acquire registry data on MipAC readmissions, hospital admissions, and mortality after one year.

The investigators will recruit 1-4 MipAC physicians to take part in the study. The project physicians will be responsible for the patient's general medical treatment, but will also perform a structured, clinical drug review that goes beyond what is considered usual care. The project physicians will provide necessary information on the patient's medical history and drug use from the medical records, carry out a medical history from the patient, and a physical examination. Relevant blood analyses and other supplementary tests will be ordered if not already available. The clinical drug review will be aimed at evaluating whether current medications are indicated, whether the patient's medical conditions are satisfactorily compensated, whether dosages are appropriate, whether the patient has adverse drug effects, and whether drug-drug or drug-disease interactions are present or likely to occur. The investigators will develop a structured framework for the drug reviews, and the MipAC physicians will receive clinical supervision from a consultant in geriatric medicine.

After performing the clinical drug review, the MipAC physician will offer the patient's FP a telephone based or digital meeting with the purpose of combining the assessments of the MipAC physician and the competence of the FP in a common drug review. The two physicians will review the patient's drug list systematically and discuss if any adjustments should be done, as well as the patient's need for further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 70+
* Admitted to the MipAC unit
* Use of at least six different systemic medications taken regularly
* Informed consent by the patient

Exclusion Criteria:

* Previously included in the study
* Not speaking or understanding Norwegian
* Residing outside of the municipality of Oslo
* Planned discharge within 24 hours
* Isolated for infection control reasons
* Considered too ill to approach or life expectancy judged to be less than six months
* Personnel at the MipAC unit discourage participation (in case of important reasons not covered by the other exclusion criteria)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 139 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) | 16 weeks
  HRQoL assessed with the 15-dimensional instrument 15D. 15D is a generic, 15-dimensional instrument concerning different aspects of HRQoL. The dimensions are mobility, vision, hearing, breathing, sleeping, eating, speech, elimination, usual activities, mental function, discomfort and symptoms, depression, distress, vitality, and sexual activity. Each dimension is rated on an ordinal scale with five levels, and the respondent chooses the level best describing his/her present health status. Single index scores are calculated by population-based utility weights, and range from 0 to 1, with higher scores indicating better HRQoL.

SECONDARY OUTCOMES:
Handgrip strength | 16 weeks
  Handgrip strength measured with a standard dynamometer, with three attempts on each hand. The highest value of all six attempts will be reported, measured in kilograms.
Digit span forward | 16 weeks
  Results will be reported as the maximum digit span completed.
Digit span backwards | 16 weeks
  Results will be reported as the maximum digit span completed.
Unstimulated whole saliva flow | 16 weeks
  Unstimulated whole saliva flow will be measured by the spitting method by weighing plastic cups before and after a collection period of 3 minutes. Results will be reported as milliliters/minute.
The Shortened Xerostomia Inventory (SXI) | 16 weeks
  The Shortened Xerostomia Inventory (SXI) is a five-item summated rating scale which combines the responses to five individual items into a single sum score. The sum score can range from 5 to 15, with higher values representing more severe xerostomia.
The eight-item Visual Analog Scale xerostomia questionnaire | 16 weeks
  This is a Visual Analog Scale with eight questions related to xerostomia where participants will be asked to mark their response to each item by placing a vertical line on the 100 millimeter horizontal scale. Results will be reported as millimeters.
Oral pain/discomfort | 16 weeks
  The patients will be asked if they have experienced any oral pain/discomfort since the KAD stay. Responses will be given on a five-category rating scale ranging from "never" (0), "hardly ever" (1), "occasionally" (2), "often" (3), to "very often" (4).
Orthostatic blood pressure | 16 weeks
  Supine blood pressure and pulse rate will be measured after a minimum of five minutes of rest. The patient will then stand up, and measurements will be repeated after one and three minutes. Orthostatic hypotension will be defined as a fall in systolic blood pressure of at least 20 mmHg or a fall in diastolic blood pressure of at least 10 mmHg after one and/or three minutes in standing position.
Falls | 16 weeks
  Number of falls.
Admissions to health institutions | 16 weeks and 1 year
  The combined number of hospital admissions and MipAC readmissions in the period from baseline to week 16. We also plan to acquire these data after one year.
Mortality | 16 weeks and 1 year
  Mortality in the period from baseline to week 16. We also plan to assess mortality after one year.

OTHER OUTCOMES:
Environmental impact measures | 16 weeks
  Environmental impact analysis will follow life cycle assessment according to the International Organization for Standardization (14040) standards to quantify greenhouse gas emissions. We will include data such as types and quantities of medications administered, types and quantities of medical equipment used during the KAD stay, number and length of hospital admissions, nursing home admissions and KAD readmissions, and number of outpatient and FP consultations.
  These data will be assessed and converted to carbon dioxide equivalents, and combined to report the environmental impact of the intervention expressed in carbon dioxide equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Romskaug, MD, PhD, Principal Investigator — Dept. of Geriatric Medicine, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 9 months and ending 3 years following publication of the main results of the study.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. As for now, we plan to upload data to Sikt (www.sikt.no) or a similar service for depositing and sharing data.

REFERENCES:
- [Derived] Santervas LR, Wyller TB, Skovlund E, Jensen JL, Fjeld KG, Hove LH, Ringstad IB, Nordberg LB, Mellingen KM, Kristoffersen ES, Romskaug R. Cooperation across healthcare service levels for medication reviews in older people with polypharmacy admitted to a municipal in-patient acute care unit (The COOP II Study): study protocol for a randomized controlled trial. Trials. 2024 Sep 13;25(1):612. doi: 10.1186/s13063-024-08442-w. PMID 39272164